CLINICAL TRIAL: NCT00651807
Title: Phase II, Randomized, Double-Blind, Placebo-Controlled Trial Investigating the Efficacy and Safety of Org 3236 Tablets in Men With Lower Urinary Tract Symptoms (LUTS) Suggestive of Benign Prostatic Hyperplasia (BPH)
Brief Title: A Trial to Investigate the Effectiveness and Safety of Org 3236 (Etonogestrel) Tablets in Men With Urinary Complaints Suggestive of a Benign Enlargement of the Prostate (304001)(P05806)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P05806; 304001
Record Dates: First submitted 2008-03-31; First posted 2008-04-03 (Estimated); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Benign Prostatic Hyperplasia (BPH)
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — etonogestrel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator): etonogestrel
  Interventions: Drug: etonogestrel
- Arm 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: etonogestrel — Lowest dose of Org 3236 per two days, lowest dose of Org 3236 per day, highest dose of Org 3236 per day for 8 weeks
  Other Names: Org 3236
  Arms: Arm 1
Drug: Placebo — Every day one tablet up to 8 weeks
  Arms: Arm 2

SUMMARY:
This trial is conducted to evaluate the effect of etonogestrel in comparison to placebo on:

* the prostate volume and the urinary complaints;
* the urinary flow and the urinary volume in the bladder after voiding;
* the progression of the disease;
* the sexual function, well-being and urinary complaints-related Quality of Life. In addition the safety and the way the drug is absorbed and excreted by the body will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent, obtained before screening evaluations;
* Men diagnosed with LUTS suggestive of BPH: Baseline IPSS score of = 12 (moderate to severe); Prostate volume of = 40 mL and < 100 mL (based on TRUS); Peak urinary flow rate = 15 mL/s with a voided volume of =125 mL
* Age at least 50 but not older than 80 years at screening
* PSA < 10 ng/mL and exclusion of prostate cancer to the satisfaction of the investigator (e.g. by biopsy)

Exclusion Criteria:

* A post void residual volume >250 mL
* Use of drugs interfering with efficacy assessments within two weeks or six months prior to start treatment (depending on drug)
* Acute urinary retention within the past 12 months
* History of surgery for BPH, including other minimally invasive procedures
* Presence of urinary tract infection
* Presence or history of (subclinical) prostate cancer, bladder cancer, urethral stricture, or pelvic irradiation
* Cardiac or cerebrovascular event within the past six months
* Presence or history of any neurological disease associated with primary bladder dysfunction
* Presence or history of liver/renal disease or disturbance of liver/renal function that failed to return to normal
* Clinically relevant abnormal laboratory result as judged by the (sub)investigator

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
The effect of Org 3236 on prostate volume compared to placebo | Screening (days -30 to -1), weeks 8, 12 and 24
The effect of Org 3236 on LUTS compared to placebo | Screening up to and including week 24
The effect of Org 3236 on urinary flow and postvoid residual volume compared to placebo | Screening and weeks 2 - 24
The effect on progression of LUTS | Screening up to and including week 24
The effect of Org 3236 on sexual function; well-being and LUTS-related Quality of Life compared to placebo | Screening and weeks 4 - 24; screening and weeks 2 - 24, respectively
The safety of Org 3236 | Screening up to and including week 24
The pharmacokinetic (Org 3236) and pharmacodynamic (T, DHT, LH, FSH, E2, SHBG) properties | Randomization and weeks 2 - 8; randomization and weeks 2 - 12 and 24, respectively

REFERENCES:
- [Background] Madersbacher S, Alivizatos G, Nordling J, Sanz CR, Emberton M, de la Rosette JJ. EAU 2004 guidelines on assessment, therapy and follow-up of men with lower urinary tract symptoms suggestive of benign prostatic obstruction (BPH guidelines). Eur Urol. 2004 Nov;46(5):547-54. doi: 10.1016/j.eururo.2004.07.016. PMID 15474261
- [Background] Gonzalez CM, McVary KT. The role of combination therapy for lower urinary tract symptoms secondary to benign prostatic hyperplasia. Curr Urol Rep. 2003 Aug;4(4):276-81. doi: 10.1007/s11934-003-0084-1. No abstract available. PMID 12882718
- [Background] McConnell J, Abrams P, Denis L, Khoury S, Roehrborn C (eds). Male Lower Urinary Tract Dysfunction - Evaluation and Management. Edition 2006 Paris, France: Editions 21, ISBN 0-9546956-6-6.